CLINICAL TRIAL: NCT07068958
Title: A Phase 2, Multi-center, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy and Safety of RCI001 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye
Brief Title: A Study Evaluating the Efficacy and Safety of RCI001 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDC001_201
Record Dates: First submitted 2025-06-27; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.25% RCI001 Ophthalmic Solution BID (Experimental): 0.25% RCI001 Ophthalmic Solution BID
  Interventions: Drug: 0.25% RCI001 Ophthalmic Solution
- Placebo Ophthalmic Solution BID (Placebo Comparator): Placebo Ophthalmic Solution (vehicle) BID
  Interventions: Drug: Placebo Ophthalmic Solution (vehicle)
- 0.25% RCI001 Ophthalmic Solution QID (Experimental): 0.25% RCI001 Ophthalmic Solution QID
  Interventions: Drug: 0.25% RCI001 Ophthalmic Solution
- Placebo Ophthalmic Solution QID (Placebo Comparator): Placebo Ophthalmic Solution (vehicle) QID
  Interventions: Drug: Placebo Ophthalmic Solution (vehicle)

INTERVENTIONS:
Drug: 0.25% RCI001 Ophthalmic Solution — 0.25% RCI001 Ophthalmic Solution
  Arms: 0.25% RCI001 Ophthalmic Solution BID; 0.25% RCI001 Ophthalmic Solution QID
Drug: Placebo Ophthalmic Solution (vehicle) — Placebo Ophthalmic Solution (vehicle)
  Arms: Placebo Ophthalmic Solution BID; Placebo Ophthalmic Solution QID

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of 0.25% RCI001 Ophthalmic Solution twice a day (BID) and four times a day (QID) compared to placebo (vehicle) in the treatment of the signs and symptoms of dry eye.

The secondary objective of this study is to evaluate the optimal dosing frequency of 0.25% RCI001 Ophthalmic Solution (BID versus QID) in the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be at least 18 years of age at the Screening Visit (Visit 1), of either gender and any race; 2. Provide written informed consent; 3. Be willing and able to comply with all study procedures; 4. Have a patient-reported history of dry eye for at least 6 months prior to Visit l; 5. Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit l; 6. Have a best corrected visual acuity (BCVA) of 0.7 logarithm of the minimum angle of resolution (logMAR) or better (Snellen equivalent score of 20/100 or better) in each eye at Visit l; 7. Report a score of ≥ 3 according to the Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire in at least one of the dry eye symptoms at Visits 1 and 2; 8. Have a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2; 9. Have a total corneal fluorescein staining score of ≥ 6 and an inferior region score of ≥ 2 (in the same eye) according to the Ora Calibra® Corneal and Conjunctival Staining Scale in at least in at least one eye at Visits 1 and 2 pre-CAE®; 10. Have a total conjunctival lissamine green staining score of ≥ 2; 11. Have a conjunctival redness score ≥ 1 according to the Ora Calibra® Conjunctival Redness for Dry Eye Scale in at least one eye at Visits 1 and 2 pre-CAE®; 12. Demonstrate in the same eye(s) a response to the CAE® at Visits 1 and 2 as defined by:

  1. Having at least a ≥ 1 point increase in fluorescein staining in the inferior region in at least one eye following CAE® exposure;
  2. Reporting an Ocular Discomfort score ≥ 3 at 2 or more consecutive time points in at least one eye during CAE® exposure (if a subject has an Ocular Discomfort rating of 3 at time = 0 for an eye, s/he must report an Ocular Discomfort rating of 4 for two consecutive measurements for that eye). Note: a subject cannot have an Ocular Discomfort score of 4 at time = 0); 13. Have at least one eye, the same eye, satisfy all criteria for 8, 9, 10, 11 and 12 above; 14. A negative urine pregnancy test if female of childbearing potential (those who are not surgically sterilized [bilateral tubal ligation, hysterectomy or bilateral oophorectomy] or post-menopausal [12 months after last menses]) and must use adequate birth control through the study period. For non-sexually active females, abstinence may be regarded as an adequate method of birth control.

Exclusion Criteria:

* 1. Have any clinically significant slit lamp findings at Visit l that may include active blepharitis, meibomian gland dysfunction, severe lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters; Note: Patients with moderate to severe meibomian gland dysfunction, in the opinion of the investigator, will not be eligible to participate in the study.

  2. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit l; 3. Have worn contact lenses within 7 days of Visit l or anticipate using contact lenses during the study; 4. Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last l2 months; 5. Have used Restasis®, Xiidra®, Cequa®, Eysuvis®, or Tyrvaya®, Vevye® within 45 days of Visit l; 6. Have had any ocular and/or lid surgeries in the past 6 months or have any planned ocular and/or lid surgeries over the study period; 7. Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit l; 8. Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study); the respective wash-out periods are required for the following medications: Confidential 6
  1. Antihistamines (including ocular): 72 hours prior to Visit 1
  2. Oral aspirin or aspirin-containing products allowed if dose has been stable over past 30 days prior to Visit 1 and no change in dose is anticipated during the study period
  3. Corticosteroids or mast cell stabilizers (including ocular): l4 days prior to Visit 1
  4. Any medication (oral or topical) known to cause ocular drying that has not been administered as a stable dose for at least 30 days prior to Visit 1 and during the study
  5. All other topical ophthalmic preparations (including artificial tear substitutes) other than the study drops: 72 hours prior to Visit 1 9. Have an uncontrolled systemic disease 10. Be a woman who is pregnant, nursing, or planning a pregnancy; 11. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 4 (or early termination visit) if of childbearing potential. Non-childbearing potential is defined as a woman who is permanently sterilized (e.g., has had a hysterectomy or tubal ligation), or is post- menopausal (without menses for l2 consecutive months); 12. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; intrauterine device; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study; 13. Have a known allergy and/or sensitivity to the test article or its components; 14. Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study; 15. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1; 16. Be unable or unwilling to follow instructions, including participation in all study assessments and visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Corneal staining sign measured with the Ora Calibra® Corneal and Conjunctival Staining Scale, and Ocular Discomfort symptom measured with Ora Calibra® Ocular Discomfort Scale in subjects dosed with 0.25% RCI001 Ophthalmic Solution BID, QID or Placebo | 4 weeks
  The objective of this study is to evaluate the safety and efficacy of 0.25% RCI001 Ophthalmic Solution twice a day (BID) and four times a day (QID) compared to placebo (vehicle) in the treatment of the signs and symptoms of dry eye

SECONDARY OUTCOMES:
Determine dosing frequency for subjects using the Ora Calibra® Corneal and Conjunctival Staining Scale for Grading of Fluorescein Staining, Ocular Surface and Disease Index (OSDI)© for Dry Eye, and Ora Calibra® Ocular Discomfort Scale for Dry Eye scores. | 4 weeks
  The secondary objective of this study is to evaluate the optimal dosing frequency of 0.25% RCI001 Ophthalmic Solution (BID versus QID) in the treatment of the signs and symptoms of dry eye.